CLINICAL TRIAL: NCT06365697
Title: Efficacy and Safety of the Ton-bridge Carotid Stent for the Treatment of Carotid Artery Stenosis: a Prospective, Multicenter, Non-inferiority, Randomized Controlled Trial
Brief Title: Evaluation of the Ton-bridge Carotid Stent for Carotid Artery Stenosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ton-Bridge Medical Tech. Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZHTQ202301
Record Dates: First submitted 2024-04-09; First posted 2024-04-15 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Carotid Artery Stenosis
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Carotid artery stenting with the experimental device
  Interventions: Device: Ton-bridge carotid stent
- control group (Active Comparator): Carotid artery stenting with the control device
  Interventions: Device: WALLSTENT carotid stent

INTERVENTIONS:
Device: Ton-bridge carotid stent — carotid artery stenting with Ton-bridge carotid stent
  Arms: experimental group
Device: WALLSTENT carotid stent — carotid artery stenting with WALLSTENT carotid stent
  Arms: control group

SUMMARY:
The purpose of this trial is to evaluate effectiveness and safety of the Ton-bridge carotid stent for the treatment of carotid artery stenosis.

DETAILED DESCRIPTION:
This is a prospective, multicenter, open-label, non-inferiority, randomized controlled trial carried out in 7 research centers in China. Patients with carotid atherosclerotic stenosis will be randomized (1:1) to either the Ton-bridge carotid stent or WALLSTENT carotid stent for treatment. The purpose of this clinical trial is to evaluate the effectiveness and safety of a novel carotid stent, the Ton-bridge carotid stent, in humans for treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18-80 years old and of any sex;
* Patient is diagnosed with carotid atherosclerotic stenosis by imaging. The lesion site is located in the extracranial segment of carotid artery and is suitable for endovascular treatment. Patient is either symptomatic with carotid stenosis≥50% or asymptomatic with carotid stenosis≥70% as determined by digital subtraction angiography (DSA) using NASCET methodology.

  * Symptomatic is defined as non-disabling ischemic stroke (mRS≤2) or transient cerebral ischemia (TIA, including cerebral hemispheric neurological events and amaurosis fugax) associated with the carotid stenosis within the past 6 months.
* The target vessel reference diameter ranges from 3.5mm to 9mm.
* Patient has been informed of the nature of this trial, understood the purpose of this clinical investigation, and volunteered to participate and sign the informed consent form.

Exclusion Criteria:

* Evolving stroke within 3 months before index procedure, disabling stroke (mRS≥3) before the procedure, or massive cerebral infarction (area of infarction is >1/3 of the ipsilateral middle cerebral artery territory) within 30 days before the procedure.
* Myocardial infarction within 30 days prior to index procedure.
* Severe heart, lung, liver, or renal insufficiency.
* Patient has known bleeding diathesis, or contraindication to heparin or antiplatelet therapy.
* Patient has a known allergy to contrast media or nickel-titanium material.
* Disturbance of consciousness, dementia, or severe neurological deficits (NIHSS≥15 or mRS≥3)
* Severe hypertension (Systolic blood pressure≥180mmHg and/or diastolic blood pressure≥110mmHg) difficult to be controlled.
* Patient has known risk factors for embolization.
* Patient has had any major surgical procedure (i.e., intraabdominal or intrathoracic surgery, any surgery or interventional procedure involving cardiac, cerebral or vascular system) within 30 days before index procedure.
* Patient has had any intracranial surgery or intracranial hemorrhage within 1 year before index procedure.
* Patient has other known neurological diseases such as intracranial tumor, which may confound the neurological assessments.
* Intracranial aneurysm or arteriovenous malformation, which requires treatment.
* Patient has other known vascular lesion requiring intervention at the same time or within 30 days after index procedure.
* Patient has other carotid diseases such as vasculitis, carotid dissection, carotid aneurysm and fibromuscular dysplasia.
* Ipsilateral intracranial artery severe stenosis (≥70%), occlusion or dissection; stenosis(≥50%) or occlusion of ipsilateral common carotid artery opening or brachiocephalic artery; any previously placed stent in the ipsilateral carotid artery or brachiocephalic artery; the target lesion is a restenosis after a previous carotid endarterectomy (CEA).
* The target lesion vessel has intraluminal filling defect, thrombosis, occlusion or subtotal occlusion ("string sign").
* Severe tortuous anatomy or other anatomic factors that prohibit the safe placement of the catheter or stent systems.
* Pregnant or lactating female.
* Patient is participating in an investigational drug or device study where the primary endpoint has not yet been completed or that will clinically interfere with the endpoint of this investigation.
* Other circumstances which the investigator considers unsuitable for participating in this investigation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of non-MAE(major adverse events) within 30 days post-procedure | Up to 30 days
  MAE is defined as any death, stroke or myocardial infarction.

SECONDARY OUTCOMES:
Technical success | Intraprocedure
  Proportion of participants who achieve technical success. Technical success is defined as successful implantation of the carotid stent and successful retraction of the delivery catheter.
Procedural success | before discharge or up to 7 days
  Proportion of participants who achieve procedural success. Procedural success is defined as stent technical success with <50% residual stenosis and no MAE in-hospital or 7 days post-procedure.
Target lesion revascularization (TLR) rate | Up to 1 year
  TLR is defined as any invasive revascularization procedure that is performed to reperfuse or increase the luminal diameter of the vessel inside or within 5mm of the previously treated lesion.
Ipsilateral stroke between 31 days and 1 year post-procedure | Between 31 days and 1 year
  Incidence of any ipsilateral stroke between 31 days and 1 year post-procedure.
In-stent restenosis rate | 180±30 days, 360±30 days
  In-stent restenosis is defined as ≥50% diameter stenosis within the stented lesion or within 5mm proximal or distal to the stent.
mRS score | 30±7 days, 180±30 days, 360±30 days
  Modified Rankin Scale (mRS) score of participants in every evaluation time point. The mRS score is generally to assess disability in patients who have suffered a stroke and ranges from 0 to 6. Higher scores mean a more severe disability. 6 means death.
Device deficiency | Up to 1 year
  Defined as the unreasonable risk that may endanger human health and life safety in the normal use of medical devices during clinical investigations, such as labeling errors, quality problems, malfunctions, etc.
Incidence of MAE | Up to 1 year
  MAE is defined as any death, stroke or myocardial infarction.
Incidence of Adverse events (AE) | Up to 1 year
  Defined as untoward medical event occurring during the course of clinical investigation, whether or not related to the medical device.
Incidence of Serious adverse events (SAE) | Up to 1 year
  Defined as the event occurring during the course of clinical investigation, which leads to death or serious deterioration in the health, including a life-threatening illness or injury; a permanent impairment of a body structure or a body function; in-patient or prolonged hospitalization; medical or surgical intervention to prevent permanent impairment to a body structure or a body function; foetal distress, foetal death, congenital abnormality or birth defect, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Liqun Jiao, Principal Investigator — Central Hospital Affiliated to Shangdong First Medical University; Yong Zhang, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (7):
- China (7):
  - The People's Hospital of Liaoning Province, Shenyang, Liaoning
  - Linyi People's Hospital, Linyi, Shandong
  - Qingdao Central Hospital, Qingdao, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Central Hospital Affiliated to Shangdong First Medical University, Jinan, Shangdong
  - Lishui Central Hospital, Lishui, Zhejiang
  - Xuanwu Hospital, Capital Medical University, Beijing